CLINICAL TRIAL: NCT07111780
Title: The Effect of Coordinative-Based Physical Activity Practices on Motor Competence, Cognitive Function and Mood in Adolescents
Brief Title: Physical Activity on Motor Competence, Cognitive Function and Mood in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Namik Kemal University (Other)
Collaborators: Princess Nourah Bint Abdulrahman University (Other)
Responsible Party: Principal Investigator, umut canlı, Prof. Dr., Namik Kemal University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2023.165.09.15
Record Dates: First submitted 2025-07-15; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Healthy; Adolescent
Keywords: motor coordination; executive function; inhibition
MeSH Terms: conditions — Inhibition, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Coordinative-Based Physical Activity Practices"program (Experimental): "Coordinative-Based Physical Activity Practices" program training group
  Interventions: Other: "Coordinative-Based Physical Activity Practices" training group
- Control group (No Intervention): Control group: The control group continued to attend standard physical education classes. In addition, the control group was not allowed to participate in any physical activity program during the study period

INTERVENTIONS:
Other: "Coordinative-Based Physical Activity Practices" training group — In the first session, participants were asked to fill in an information form, including demographic information. They were asked to complete the Brunel Mood Scale and the International Physical Activity Questionnaire (IPAQ). participants' height and body weight were measured. Participants' height was measured with a portable statiometer. Body weight was measured with a digital scale witha precision of 0.1 kg. In the second session, Go/No-Go and mental rotation tests, which are used to evaluate the cognitive functions of the participants, were administered to the participants. The KTK3+ motor competence test was used to determine the motor competence of the participants.The tests were administered to the participants in the same order and by the same researchers. Before the assessment of KTK3+ test of 5 minutes of running and 5 minutes of dynamic stretching was performed. Coordination-based physical activity applied to the exercise group continued for 25-30 minutes twice for 8 weeks.
  Other Names: Coordinative-Based Physical Activity Practices" program training group
  Arms: "Coordinative-Based Physical Activity Practices"program

SUMMARY:
The study aimed to determine the effect of coordinative-based physical activity practices on motor competence, cognitive function and mood levels of adolescent boys. It is thought to answer the questions about the effect of coordinative-based physical activity programs on motor competence, cognitive functions and mood in adolescent males and the level of this effect.

DETAILED DESCRIPTION:
The study aimed to determine the effect of coordinative-based physical activity practices on motor competence, cognitive function, and mood levels of adolescent boys. The research group consisted of 40 volunteer male students (age = 14.38±0.40) studying in a public high school. After the baseline assessment, participants were randomly divided into training (TG; n=20) or control (CG; n=20) groups in a 1:1 ratio. The physical activity levels of the participants were determined using the International Physical Activity Questionnaire (IPAQ). The KTK3+ test battery was used to determine the level of motor competence. In the evaluation of cognitive functions, the Go/No-Go test was used to measure inhibition control, and the Mental Rotation test was used for spatial-spatial cognition. The Brunel Mood Scale was used to determine the mood level of the participants.

ELIGIBILITY:
Inclusion Criteria:

* Typically developing children
* Aged between 14 and 15 years
* Enrolled in the 9th grade of high school
* Not currently taking any medication
* Provided informed consent from both the child and their parent/guardian

Exclusion Criteria:

* Having any diagnosed cardiovascular, neurological, orthopedic, or psychiatric condition
* Taking regular medication
* Outside the age range of 14-15 years
* Presence of any developmental disorder or learning disability

Ages: 14 Years to 15 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2024-04-15 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-07-05 (Actual)

PRIMARY OUTCOMES:
Changes in motor competence performance (KTK3+ Test Batery) | before and at the end of the 8-week intervention
  The KTK3+ test battery, supported by a hand-eye coordination task, was used to assess children's motor competence. It is determined that KTK3+ test was a highly valid and reliable measurement tool to be used by Turkish children. KTK3 measures general gross motor coordination. By adding a throwing and catching task to the KTK3 test form, the KTK3+ test battery covering three fundamental motor skill domains (movement, balance, and object control) was developed. The KTK3+ test includes balancing backwards (BB), moving sideways (MS), jumping sideways (JS), and hand-eye coordination task (EHC).
Changes in inhibitory control (Go/no-go test) | before and at the end of the 8-week intervention.
  The Go/No-Go test is the most widely used in inhibitory control assessment. In this study, a computer-based Go/No-Go test was applied. The test consists of five sections in total. Each section consists of 40 trials and each section contains 20 X (go) stimuli and 20 O (no-go) stimuli. A rest period of 10 seconds was given between the sections. There were 100 X (go) and 100 O (no-go) stimuli in total. These stimuli are displayed on the screen for 50 milliseconds and then there is a black screen for 1450 milliseconds.
Changes in mental rotation (Mental Rotation Test) | before and at the end of the 8-week intervention.
  Mental rotation is defined as the ability to visualize the position and movement of a two- or three-dimensional object in space. As a result of neuroimaging studies showing that mental rotation and movement readiness may have common mechanisms in the premotor cortex, it has been suggested that there is a link between mental rotation test performance and physical activity. In this study, a computer-based mental rotation test was used. The test consists of a total of 16 trials. There are four images on the screen and these images are created by adding 10 cubes end to end. While the image on the left is the reference, only one of the other three images is a rotated view of the reference image in 3D space. The other two images are mirror images of the reference image. The correct answers in the first eight questions were rotated on the X axis and the correct answers in the other eight questions were rotated on the Z axis.
Changes in mood (Brunel Mood Scale) | before and at the end of the 8-week intervention
  Brunel mood scale was developed by Terry and colleagues. The scale was adapted into Turkish by Soylu and colleagues. The scale consists of six (6) sub-dimensions and 24 items. In the adapted study, internal consistency was reported as α=.83 for the anger subscale, α=.81 for the confusion subscale, α=.81 for the depression subscale, α=.81 for the fatigue subscale, α=.88 for the tension subscale and α=.75 for the vitality subscale. In the current study, α=.76 for the anger subscale, α=.73 for the confusion subscale, α=.77 for the depression subscale, α=.83 for the fatigue subscale, α=.82 for the tension subscale and α=.80 for the vitality subscale.High scores on the scale indicate a high mood value.

CONTACTS AND LOCATIONS:
Overall Officials: selim esgiyayla, Study Director — depatment of physical education and sport
Locations (1):
- Namık Kemal, Tekirdağ, süleymanpaşa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The sample group consists of adolescent children under the age of 18. In the voluntary participant and parent form, it is stated that the data of the participants will not be shared with third parties.

REFERENCES:
- [Background] Rodriguez-Ayllon M, Cadenas-Sanchez C, Estevez-Lopez F, Munoz NE, Mora-Gonzalez J, Migueles JH, Molina-Garcia P, Henriksson H, Mena-Molina A, Martinez-Vizcaino V, Catena A, Lof M, Erickson KI, Lubans DR, Ortega FB, Esteban-Cornejo I. Role of Physical Activity and Sedentary Behavior in the Mental Health of Preschoolers, Children and Adolescents: A Systematic Review and Meta-Analysis. Sports Med. 2019 Sep;49(9):1383-1410. doi: 10.1007/s40279-019-01099-5. PMID 30993594
- See also: protocol — https://pubmed.ncbi.nlm.nih.gov/30993594/
- Available data/document: Study Protocol: example study protokol — https://www.nature.com/articles/s41598-024-79811-3